CLINICAL TRIAL: NCT04729192
Title: Translation and Validation of the Turkish Version of the ObsQoR-10 Questionnaire (ObsQoR-10T)
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Other Study IDs: ObsQoR-10T
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Quality of Recovery; Delivery
Keywords: ObsQoR-10T Questionnaire

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: The patients will complete the ObsQoR-10T questionnaire on day 1 following delivery
  Interventions: Other: ObsQoR-10T Questionnaire

INTERVENTIONS:
Other: ObsQoR-10T Questionnaire — The ObsQoR-10T questionnaire consists of 10 items assessing physical comfort and pain, physical independence, and emotional status. Each item is scored from 0 to 10 and the total score is the sum of the score for each item, which is a score from 0 to 110.

SUMMARY:
The quality of recovery scoring tools for the obstetric patient population is limited. In 2019, Ciechanowicz et al. developed and validated a postpartum recovery score; the ObsQoR-11; used following elective and non-elective cesarean delivery. The ObsQoR-11 was modified to the ObsQoR-10 by Sultan et al. and used spontaneous and operative vaginal delivery based on patient feedback. There is currently only a Hebrew version of this recovery score. ObsQoR has not yet been validated for use in Turkish, which is one of the most spoken languages in the World. Therefore the investigators aimed to psychometrically evaluate (assess validity, reliability, and clinical feasibility) the Turkish translated version of the ObsQoR-10 PROM in a Turkish cohort of women.

ELIGIBILITY:
Inclusion Criteria:

* Turkish-speaking women (in Turkey) greater than 18 years of age who are also able to read and understand written Turkish
* Spontaneous vaginal delivery with or without neuraxial anesthesia for labor analgesia (including repair of vaginal tears and manual removal of the placenta) or elective cesarean delivery
* Women who have singleton births
* Primiparous (first baby) -≥38 weeks gestational age

Exclusion Criteria:

* Psychiatric or neurological pathology compromising cooperation in the questionnaire validation protocol,
* Age < 18 years
* Women whose infants have died
* Mother or baby requiring ICU after delivery.
* Patient refusal to participate
* Inability to read or understand written Turkish
* Failed neuraxial analgesia: elective cesarean delivery
* General anesthesia
* Intrapartum cesarean
* Assisted/operative (i.e. vacuum, forceps) vaginal delivery

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: All patients admitted for spontaneous obstetrical labor or scheduled cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Validity of Obstetric Quality of Recovery-10 Turkish (ObsQoR-10T) questionnaire | on day 1 following delivery
  Evaluate the validity of the Turkish version of the ObsQoR-10 to assess immediate postpartum recovery following vaginal delivery or Caesarean section.The ObsQoR-10 based on patient feedback regarding the 0-10 scoring for "negative symptoms" such as pain, nausea and vomiting and dizziness (found in questions 1-4 of ObsQoR- 10) and "positive" symptoms such as comfort and feeling in control (found in questions 5-10 of ObsQoR-10). Overall higher recovery scores indicate better recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Betul Kozanhan, Konya, Turkey (Türkiye)